CLINICAL TRIAL: NCT05290831
Title: Changes in Heart Rate Variability And Heart Rate/Activity Slope Measures After Hospitalization for Acute Exacerbations of COPD: An Observational Study
Brief Title: Changes in Heart Rate Variability And Heart Rate/Activity Slope After Hospitalization for Acute Exacerbations of COPD
Acronym: CHARM COPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minneapolis Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, David MacDonald, Principal Investigator, Minneapolis Veterans Affairs Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1653926
Record Dates: First submitted 2022-03-11; First posted 2022-03-22 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Main study group (Experimental)
  Interventions: Device: VitalPatch

INTERVENTIONS:
Device: VitalPatch — The VitalPatch continuously monitors skin temperature, activity, and electrocardiography.

SUMMARY:
The purpose of this study is to observe the variation in time between heart beats and how heart rate changes during activity evolve after hospitalization for an exacerbation of COPD.

DETAILED DESCRIPTION:
The investigators will place a monitoring patch that continuously records electrocardiogram and activity. Participants will switch this patch every 7 days for a total of 28 days. From these data the investigators will observe how heart rate variability and heart rate responses to exercise evolve after hospitalization for an exacerbation of COPD.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. At least moderate COPD by Global Initiative for Chronic Obstructive Lung Disease spirometry criteria (FEV1/FVC < 0.7 and FEV1 < 80% predicted)
3. 10 pack year smoking history
4. Hospitalized with one or more of:

   1. increased dyspnea
   2. increased sputum
   3. change in sputum character
5. Treated with corticosteroids and/or antibiotics for respiratory indications
6. Age > 40 years old

Exclusion Criteria:

1. Discharging home on hospice
2. Inability to follow trial protocols
3. Pacemaker
4. Allergy to a component of the adhesive patches
5. Breastfeeding
6. Permanent/continuous atrial fibrillation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2022-04-10 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Model fit from repeated measures mixed model of heart rate/activity slope | 28 days
  The investigators will average heart rate and activity (from accelerometer output) over 30-second periods. The highest 30-second average from each 5 minute period will be used to create the heart rate/activity slope for each 24-hour period while the device is worn. They will then model the change in heart rate/activity slope using a linear-mixed effect model with a random intercept and slope for each individual.
Heart rate variability slopes (time and frequency-domain) | 28 days
  The investigators will use Kubios software to calculate heart rate variability (time and frequency domain measurements) for each 24-hour period that the patch is worn. They will use repeated mixed measures models with random intercept and slope to model the change in heart rate variability after discharge.

SECONDARY OUTCOMES:
Comparison of heart rate/activity slope in participants readmitted vs not-readmitted | 28 days
  The investigators will compare heart rate/activity slope in participants who are readmitted to the hospital within 28 days to those who are not readmitted to the hospital within 28 days using a linear mix-effect model with random intercept and slope.
Comparison of heart rate variability slope in participants readmitted vs not-readmitted | 28 days
  The investigators will compare heart rate variability slopes (time and frequency domain) in participants who are readmitted to the hospital within 28 days to those who are not readmitted to the hospital within 28 days using a linear mix-effect model with random intercept and slope.
Acceptability to participants | 28 days
  We will query participants if the monitoring patch would be acceptable if it were shown to improve their care for COPD.

CONTACTS AND LOCATIONS:
Overall Officials: David MacDonald, MD, MS, Principal Investigator — Minneapolis Veterans Affairs Medical Center

IPD SHARING:
Plan to Share IPD: No